CLINICAL TRIAL: NCT00955448
Title: Randomized Controlled Trial of SIS Mesh for Anterior Repair: A Pilot Study
Brief Title: Trial of Small Intestine Submucosa (SIS) Mesh for Anterior Repair: A Pilot Study
Acronym: Anterior SIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Cook Group Incorporated (Industry); Alberta Health services (Other)
Responsible Party: Principal Investigator, Dr. Sue Ross, Adjunct Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anterior SIS 300609; Ethics: E-22217
Record Dates: First submitted 2009-08-05; First posted 2009-08-10 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Anterior Pelvic Organ Prolapse
Keywords: Anterior pelvic organ prolapse; Surgical repair; Pelvic floor surgery; Randomized clinical trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIS Mesh (Cook Medical) (Experimental): Anterior prolapse repair will be reinforced using SIS mesh
  Interventions: Device: SIS mesh (Cook Medical); Procedure: Anterior prolapse repair
- No-mesh (Active Comparator): Anterior prolapse repair with no mesh reinforcement
  Interventions: Procedure: Anterior prolapse repair

INTERVENTIONS:
Device: SIS mesh (Cook Medical) — Anterior prolapse repair will be reinforced using surgical mesh made from porcine small intestine mucosa (Cook Medical)
  Arms: SIS Mesh (Cook Medical)
Procedure: Anterior prolapse repair — Anterior prolapse repair will be conducted without using mesh reinforcement

SUMMARY:
Prolapse occurs when pelvic organs drop down and cause a bulging of the tissues. An "anterior wall prolapse" occurs when the front of the vagina loses its support, and the bladder drops down and rotates into the vaginal opening. The bladder can cause a bulge out of the vagina.

One of the treatment options available is to repair the anterior wall surgically. The goals of surgery are to return the anatomy to its usual position, ensuring that all the pelvic floor organs (bladder, vagina and rectum) can function properly. The ideal surgical repair would also be long lasting.

Two surgical options are routinely performed in Calgary for repair of an anterior compartment prolapse. One option involves fixing the organs back in place using sutures. The other option uses sutures plus a mesh made of small intestine submucosa (SIS) that is already licensed for use in Canada. The SIS mesh is slowly absorbed after it is placed in the pelvic area. The investigators do not know which of these two options is the best surgical procedure. Both may have different advantages that would result in better results. This study is designed to try and find out if one of these procedures is better, and if a larger study may be needed.

ELIGIBILITY:
Inclusion Criteria:

* Women who require surgical correction for anterior compartment prolapse. (Concomitant surgery is permitted.)
* Point Ba of 0 or greater: that is a positive Ba, indicating that the prolapse is beyond the introitus, not within the vagina.
* Patient must consent to participate in the study.

Exclusion Criteria:

* Having an obliterative procedure (Lefort procedure or colpocleisis).
* Allergy to graft material.
* Immunocompromised.
* Previous anterior compartment repair.
* Are unable to understand English.
* Will be unavailable for follow-up.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Objective assessment of prolapse. "Cure" is defined as point Ba (on POP-Q) of -1 or above (i.e., more negative) | 12 months postoperatively

SECONDARY OUTCOMES:
Change in point Ba (on POP-Q) from baseline | 12 months postoperatively
Pelvic Organ Prolapse Quantification(POP-Q) stage | 12 months postoperatively
Change in POP-Q stage from baseline | 12 months postoperatively
Postoperative complications | 12 months postoperatively
Pelvic Floor Distress Inventory short form-20 (PFDI-20) | 12 months postoperatively
Pelvic Floor Impact Questionnaire short form-7 (PFIQ-7) | 12 months postoperatively
Sexual function (Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) | 12 months postoperatively
Surgical complications | Up to 6 weeks postoperatively
Satisfaction with surgical outcome | 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Magali Robert, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Result] Robert M, Girard I, Brennand E, Tang S, Birch C, Murphy M, Ross S. Absorbable mesh augmentation compared with no mesh for anterior prolapse: a randomized controlled trial. Obstet Gynecol. 2014 Feb;123(2 Pt 1):288-294. doi: 10.1097/AOG.0000000000000105. PMID 24402595